CLINICAL TRIAL: NCT03054597
Title: Novel Way to Strengthen Eye Muscle and Enhance Peripheral Vision
Brief Title: Use of Eye Exercises to Improve Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ACSEF2012JB
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Eye Strain
MeSH Terms: conditions — Asthenopia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults (Experimental): The arm consisted of adult participants who underwent:
  Circular Light Motion exercises: 4 times over 2 weeks Diagonal Light Motion exercises: 4 times over 2 weeks Peripheral Light Motion exercises: 4 times over 2 weeks
  Interventions: Device: Circular light motion; Device: Diagonal light motion; Device: Peripheral light motion; Procedure: Exercise
- Children (Experimental): The arm consisted of child participants who underwent:
  Circular Light Motion exercises: 4 times over 2 weeks Diagonal Light Motion exercises: 4 times over 2 weeks
  Interventions: Device: Circular light motion; Device: Diagonal light motion; Procedure: Exercise

INTERVENTIONS:
Device: Circular light motion — Exercise with circular light motion
Device: Diagonal light motion — Exercise with diagonal light motion
Device: Peripheral light motion — Exercise with peripheral light motion
  Arms: Adults
Procedure: Exercise

SUMMARY:
Children in the United States watch an average of twenty-eight hours of television and play around thirteen hours of video games per week. The objective of this experiment was to see if a specific eye exercises could strengthen the eye muscles and improve the peripheral vision range of children and adults.

DETAILED DESCRIPTION:
Children in the United States watch an average of twenty-eight hours of television and play around thirteen hours of video games per week. When their eyes are focused, people tend to blink their eyes less, exacerbating the problem of eye fatigue or stress. The objective of this study is to see if a novel exercise technique can increase eye muscle strength and widen peripheral vision. Experiments were conducted by asking the test subjects to follow, with their eyes, a set of blinking LED lights on 3 vision exercise devices. These LED lights were laid in circular or diagonal configurations, and programmed using a microcontroller to blink or 'move' in certain directions and at certain speeds. An endurance score, measured as total time that the test subject completed while following the blinking LED lights before his/her eyes became tired, was recorded. Nineteen test subjects aged 12-81 were asked to exercise their eyes four times over 2 weeks using the devices for as long as they could until they experienced mild eye fatigue. Endurance scores, peripheral vision, and peripheral reading ranges were assessed before and after the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Able to read English

Exclusion Criteria:

* Cannot be colorblind

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Eye Muscle Endurance | 2 weeks
  The time spent exercising prior to eye strain

SECONDARY OUTCOMES:
Peripheral Vision | 2 weeks
  The lateral degrees at which the test subject could see a blank card
Peripheral Reading Range | 2 weeks
  The lateral degrees at which the test subject could read the letters on a card

CONTACTS AND LOCATIONS:
Locations (1):
- Hopkins Junior High School, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: No